CLINICAL TRIAL: NCT02277860
Title: Gaming Console Home-Based Exercise for Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John D Lowman, PT, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F120307002
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: Exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Aerobic and strength training using the Wii Fit Plus for ≥ 30 min, ≥3 days/week, for 12 weeks, at a moderate intensity (Borg CR10 3-5).
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Aerobic and strength training using the Wii Fit for ≥ 30 min, ≥3 days/week, for 12 weeks, at a moderate intensity (Borg CR10 3-5).

SUMMARY:
Physical activity and exercise have become an accepted and valued component of cystic fibrosis care. Regular physical activity and exercise can slow the rate of decline of pulmonary function, improve physical fitness, and enhance quality of life. However, motivating people to be more active is challenging. Supervised, facility-based exercise programs are expensive and labor intensive (since groups of patients with CF cannot exercise together in the same physical location). Home-based exercise using an interactive exergame device may be an effective way to improve adherence to an exercise program for patients with CF. Therefore, the primary objective of this study is to evaluate the effects of a 12-week, home-based exergame exercise intervention on aerobic capacity (peak VO2). The secondary endpoint is nasal potential difference, an indicator of how well sodium and chloride flow across the mucous membranes in the nose. Other outcomes include patient-reported quality of life and habitual physical activity level. Following baseline assessments participants will be begin a 12 week, partially-supervised exercise program consisting of at least 90 minutes per week of aerobic and resistance exercise training using the Nintendo Wii Fit Plus exergaming device. Participants will receive at least monthly follow-up phone calls to provide additional exercise counseling and motivation. After 12 weeks, they will continue with the exergame intervention for another 12 weeks, but without external supervision.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CF
* currently sedentary (<60 min/week of physical activity)
* stable clinical condition (no exacerbation in last 6 weeks)

Exclusion Criteria:

* nasal surgery for polyposis in the past 2 years
* participating or have participated (in the past 30 days) in another clinical trial which can affect the outcomes of the proposed study
* unable to read/speak English
* recurrent pneumothorax (in the past 6 months)
* hemoptysis (hospitalized in the past 6 months)
* uncontrolled CF-related diabetes (HbA1c > 10%)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2 peak) | 12 and 24 weeks
  Measure of aerobic physical fitness

SECONDARY OUTCOMES:
Nasal potential difference (NPD) | 12 weeks
  Measure of respiratory/airway ion transport
Cystic Fibrosis Questionnaire-Revised (CFQ-R)) | 12 and 24 weeks
  Health-related quality of life questionnaire (especially respiratory-related symptoms)
Habitual physical activity level | 12 and 24 weeks
  Accelerometer-based measure of frequency, intensity and duration of bouts of physical activity while user is wearing device.

CONTACTS AND LOCATIONS:
Overall Officials: John D Lowman, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Lowman JD, Solomon GM, Rowe SM, Yuen HK. Gaming Console Home-Based Exercise for Adults with Cystic Fibrosis: Study Protocol. Int J Caring Sci. 2020 Spring/Summer;13(2):1530-1540. PMID 33163109